CLINICAL TRIAL: NCT06965673
Title: Eye-movement Dynamics During Free Viewing as a Biomarker for Assessment of Visuospatial Functions and for Closed-loop Rehabilitation in Stroke
Brief Title: Assessment of Eye Movements in Stroke Patients and Closed-loop Intervention
Acronym: EMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Collaborators: Azienda Ospedaliera di Padova (Other); University of Padova (Other)
Responsible Party: Principal Investigator, Marco Zorzi, Professor, IRCCS San Camillo, Venezia, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.09 RF-2019-12369300
Record Dates: First submitted 2025-04-23; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Visuospatial
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): This group will undergo ten sessions of the experimental visual exploration protocol and the standard neuropsychological rehabilitation delivered in the clinical facility
  Interventions: Behavioral: Visual exploration training; Behavioral: Standard neuropsychological rehabilitation
- Control (Active Comparator): This group will undergo the standard neuropsychological rehabilitation at the IRCCS San Camillo hospital
  Interventions: Behavioral: Standard neuropsychological rehabilitation

INTERVENTIONS:
Behavioral: Visual exploration training — Visual exploration of natural scenes guided by closed-loop auditory biofeedback through eye-tracking
  Arms: Intervention
Behavioral: Standard neuropsychological rehabilitation — Standard rehabilitation delivered at the IRCCS San Camillo hospital

SUMMARY:
The current study evaluates first the assumption that eye-movements during free viewing behavior are potential biomarkers of visuospatial deficits in stroke population. Second, it assesses the feasibility of a novel visual exploration training to ameliorate visuospatial deficits, by exploiting an auditory biofeedback system coupled with online parsed fixations.

DETAILED DESCRIPTION:
This study is divided into two parts concerning the diagnostic and treatment of visuospatial deficits in patients affected by unilateral stroke. Eye movements indices during free viewing of natural scenes will be correlated to the standard neuropsychological evaluation, describing the cognitive, motor and functional spectrum of patient status. Moreover, functional and structural neuroimaging will be exploited to identify neural correlates of patient eye movements characteristics. Ultimately, a subsample of randomly assigned participants, at the IRCCS San Camillo, will undergo a novel visual exploration training, in addition to the standard rehabilitation. This protocol consists of natural scene exploration guided by an auditory biofeedback system which tracks online parsed fixations. Concretely, the training maneuvers exploration toward salient regions of the presented image, as indicated by a normative sample. Changes in free viewing behavior, neuropsychological assessment and neuroimaging will be discussed compared to an active control group and a healthy sample.

ELIGIBILITY:
Inclusion Criteria:

* Vigilant
* First unifocal ischemic or hemorragic stroke
* Presence of maximum two lacunae, clinically silent, smaller than 15 mm. in the structural MRI
* Evident symptoms in the visual, attentive, memory, motor or language domain supported by the radiological exam

Exclusion Criteria:

* Previous stroke history, visible at the radiological exam
* Multifocal deficit
* Incapacity to remain vigilant during the required assessments
* Claustrophobia and/or metallic objects which could prevent MRI acquisition
* Presence of other neurological, psychiatric or medical conditions which may undermine interpretation of behavioral and neuroimaging results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change pre-post rehabilitation in eye movements patterns during free viewing | At day 0 and day 30 (i.e., end of the rehabilitation)
  Eye movements patterns described by fixations, saccades and blinks related features summarized by principal component analysis (PCA)
Change pre-post rehabilitation in Behavioral Inattention Test score | At day 0 and day 30 (i.e., end of the rehabilitation)
  Neuropsychological test assessing visuospatial deficits
Change pre-post rehabilitation in Trail Making Test score | At day 0 and day 30 (i.e., end of the rehabilitation)
  Neuropsychological test assessing visuospatial abilities, scored as the time to complete the task
Change pre-post rehabilitation in Posner Test reaction times | At day 0 and day 30 (i.e., end of the rehabilitation)
  Neuropsychological test assessing visuospatial abilities, scored with the measured reaction times
Change pre-post rehabilitation in Attention Matrices Test | At day 0 and day 30 (i.e., end of the rehabilitation)
  Neuropsychological test assessing visuospatial deficits
Change pre-post rehabilitation in Brief Visuospatial Memory Test Revised | At day 0 and day 30 (i.e., end of the rehabilitation)
  Neuropsychological test assessing visuospatial memory
Change pre-post rehabilitation in Bells Test | At day 0 and day 30 (i.e., end of the rehabilitation)
  Neuropsychological test assessing visuospatial deficits
Change pre-post rehabilitation in Apple Test score | At day 0 and day 30 (i.e., end of the rehabilitation)
  Neuropsychological test assessing visuospatial deficits
Change pre-post rehabilitation in Comb and Razor Test | At day 0 and day 30 (i.e., end of the rehabilitation)
  Neuropsychological test assessing functional activities to investigate spatial attention deficits
Change pre-post rehabilitation in Mental Number Interval Bisection | At day 0 and day 30 (i.e., end of the rehabilitation)
  Neuropsychological test investigating spatial biases in the mental number line
Change pre-post rehabilitation in Anosognosia | At day 0 and day 30 (i.e., end of the rehabilitation)
  Neuropsychological test investigating deficits awareness
Change pre-post rehabilitation in Load Test | At day 0 and day 30 (i.e., end of the rehabilitation)
  Neuropsychological test assessing spatial attentional deficits with cognitive load as a moderator
Change pre-post rehabilitation in the Catherine-Bergego Scale score | At day 0 and day 30 (i.e., end of the rehabilitation)
  Test assessing activities of daily living involving spatial attention

SECONDARY OUTCOMES:
Change pre-post rehabilitation in structural and functional connectivity | At day 0 and day 30 (i.e., end of the rehabilitation)
  Structural and functional MRI connectivity maps

CONTACTS AND LOCATIONS:
Overall Officials: Marco Zorzi, Principal Investigator — San Camillo IRCCS, Venice, Italy
Locations (2):
- Italy (2):
  - Azienda Ospedaliera di Padova, Padua, PD
  - IRCCS San Camillo, Venice-Lido, VE

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pollock A, Hazelton C, Henderson CA, Angilley J, Dhillon B, Langhorne P, Livingstone K, Munro FA, Orr H, Rowe FJ, Shahani U. Interventions for disorders of eye movement in patients with stroke. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD008389. doi: 10.1002/14651858.CD008389.pub2. PMID 21975780